CLINICAL TRIAL: NCT00571207
Title: Scientific Evaluation of Oral Fluid Screening Devices and Preceding Selection Procedures
Brief Title: Oral Fluid Screening Devices
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: KTL 402-1
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Drug-impaired Driving
Keywords: driving under the influence of drugs; on-site oral fluid screening devices; checklist

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Oral fluid and whole blood are collected. However, no DNA testing will be carried out. The research focuses on drug and medicine concentrations in these matrices.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I: Drivers suspected of driving under the influence of drugs
  Interventions: Device: On-site oral fluid screening devices; Behavioral: Checklist: drug recognition expert
- II: Drivers not suspected of driving under the influence of drugs
  Interventions: Device: On-site oral fluid screening devices; Behavioral: Checklist: drug recognition expert

INTERVENTIONS:
Device: On-site oral fluid screening devices — Comparison of screening device results to oral and/or blood sample results
Behavioral: Checklist: drug recognition expert — Correlation of drug recognition expert observations to findings for drugs in non-suspected/suspected cases

SUMMARY:
This research includes the evaluation of a checklist and on-site screening devices to pre-select drivers suspected of being drug-impaired. The reliability of a limited number of promising on-site screening devices will be investigated. The devices tested will have to be promising regarding both reliability and practicality. In addition to the scientific evaluation of the checklist and the oral fluid screening devices, the time consumption of the selection procedure as a whole (checklist + oral fluid screening) will be evaluated.

Outcome of the study will be recommendations for the roadside selection procedure of drivers suspected of drug-related impairment. The recommendations will concentrate on the reliability of the selection procedure.

The study is part of an EU project DRUID. Two other countries in Europe take part to this study along with Finland.

ELIGIBILITY:
Inclusion Criteria:

* Drivers of motorised vehicles
* 18 years or older
* Willing to participate

Exclusion Criteria:

* Younger than 18
* Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Drivers suspected of driving under the influence of drugs. Also drivers who are not suspected of driving under the influence.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-04; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
scientific evaluation of the on-site oral fluid screening devices | three years

SECONDARY OUTCOMES:
evaluation on the police checklist | three years
the time consumption of the selection procedure as a whole (checklist + oral fluid screening) | three years

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Lillsunde, Dr, Principal Investigator — National Public Health Institute
Locations (1):
- National Public Health Institute, Helsinki, Finland

REFERENCES:
- See also: Related Info — http://www.druid-project.eu